CLINICAL TRIAL: NCT07108439
Title: The Effectiveness of Intra-osseous Anaesthesia in Reducing Immediate and Delayed Post-operative Complications Associated With the Extraction of First Permanent Molars Under General Anaesthesia: A Randomised Controlled Trial
Brief Title: Usefulness of Intraosseous Anesthesia for Permanent Tooth Extraction Under GA in Pediatric Dental Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2025-0166
Record Dates: First submitted 2025-07-08; First posted 2025-08-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: No Condition, Assessment of Healthy Volunteers
Keywords: Intra-osseous anesthesia; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinding is performed using a 6 digit code generated randomly using www.random.org. This code shall be used in all the patients files and shall only be known to the trial administrator.
  It is a double blind study in which the operator knows whether she is giving intra-osseus anesthesia (articaine) or not, but the patient and the evaluator of the pre- and post- operative scales will not know if the patient got local anaesthesia or not.
  SR has the excel file with the results of the block randomisation and key for blinding (pseudonymization).
  Allocation concealment will be performed by with the sealed envelope technique.SR is independent of the study results. He has no access to the results of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra osseous administration of local anesthesia during general anesthesia (Experimental): Intra osseous administration of articain 4% 1/100 000 during general anesthesia for the extraction of a first permanent molar. The administration will be done with Quicksleeper 5.
  Interventions: Other: Administration of intra-osseous local anesthesia before the extraction of a first permanent molar under general anesthesia
- Control group (No Intervention): Normal procedure: no local anesthesia for the extraction of a first permanent molar during general anesthesia

INTERVENTIONS:
Other: Administration of intra-osseous local anesthesia before the extraction of a first permanent molar under general anesthesia — Intra osseous administration of articain 4% 1/100 000 during general anesthesia for the extraction of a first permanent molar. The administration will be done with Quicksleeper 5.
  Arms: intra osseous administration of local anesthesia during general anesthesia

SUMMARY:
The investigators are doing a study to see if a new way of giving local anesthesia during dental surgery can help children feel better after having a tooth removed under general anesthesia (when they are fully asleep). Normally, dentists give numbing medicine that can leave the lips or cheeks numb. This sometimes causes children to bite themselves without realizing it, which can make them upset when they wake up. In this study, the investigators are testing a special technique called intra-osseous anesthesia, which numbs only the tooth and not the surrounding soft tissues. The investigators hope this will reduce pain after surgery without causing numbness or accidental biting. Children in the study will be randomly placed into one of two groups: one group will receive this special anesthesia before the tooth is removed, and the other group will not. Before and after the procedure, the investigators will ask some short questions and observe the participants to check for pain, anxiety, or confusion. The parents of the participants will also receive a short online questionnaire to fill out the day after the procedure. The goal is to find out if this method helps children wake up more comfortably, feel less pain, and avoid side effects. This could improve how dentists care for children during dental treatments in the future.

DETAILED DESCRIPTION:
To investigate whether the administration of intra-osseous local anesthesia (Quicksleeper 5) to children during general anesthesia prior to the extraction of a first permanent molar has an effect on the immediate and delayed postoperative delirium, anxiety and pain in the child.

Intra-osseous anesthesia consists of 3 major steps:

1. Limited superficial anesthesia of the mucosa at the level of the tooth to be treated/extracted
2. Perforation of the bone by means of a rotating needle movement
3. Injection of the local anesthetic directly into the bone The operator (AG) will administer the intra-osseous anesthesia just before the tooth(s) are extracted. The extractions will always be performed at the end of the dental treatment.

A permanent molar must be removed from the child and this will be done under general anesthesia. Previous scientific studies have shown that when the dentist also administers local anesthesia during general anesthesia for tooth removal, children suffer from side effects of the local anesthesia. These side effects include numbness and lip or cheek biting. This can make them extra agitated when waking up from general anesthesia.

This intra-osseous anesthesia technique only anesthetizes the tooth. As a result, the child should not experience the above-mentioned side effects or to a lesser extent. In this study,The investigators want to investigate this effect. The advantage of this technique is that the child is expected to need little or no painkillers after the operation compared to the current procedure.

On the day of the procedure, upon arrival at the hospital, three short questionnaires will be administered regarding anxiety and pain. One questionnaire is observational, for the other two he investigators ask a little cooperation from the patient. This concerns the FLACC (Face, Legs, Activity, Cry, Consolability), VAS (Visual Analogue Scale) and CFSS-DS (Children's Fear Survey Schedule - Dental Scale).

If the patient is randomly assigned to the group that will receive local anaesthetic, this will be administered intra-osseously with the Quicksleeper 5 just before the tooth(s) is/are removed. The local anaesthetic that will be used is articaine 4% with epinephrine 1/100,000, this is a standard local anaesthetic in dentistry, the good and efficient effect of which has long been demonstrated.

Group 1 will receive local anaesthesia intra-osseously and group 2 will not. There is no further distinction between the groups.

The time at which the local anaesthetic is administered and the time at which the procedure is over will be noted.

After the procedure, the same questionnaires will be administered at set times as before the procedure. The patient does not have to stay in the hospital longer than normal for these questionnaires. The FLACC will be administered after 10/30/60/120 min, the VAS when the patient is able to speak and after 120 min, the CFSS-DS after 120 min and the delirium flowchart is an observational measurement that will be performed 5 min after spontaneously opening the eyes. The day after the procedure, the parents/guardian will be asked to answer one more questionnaire of approximately 20 questions via a QR code received.

ELIGIBILITY:
Inclusion Criteria:

* - Children between 6 and 12 years old, belonging to the category of ASA I or II according to the 'American Society of Anaesthesiologists'
* Children who are cooperative enough for pre- and post-operative measurements
* Children who are not allergic to components of local anaesthesia
* Children who need at least one extraction of a FPM
* Children without a hematological condition
* Children who haven't taken painkillers 48 hours before the procedure
* Patients who need a treatment under general anaesthesia (nasal intubation) due to polycaries/fear/anxiety.
* Able to obtain a written consent from the parent/guardian after explaining the full details of the treatment procedure and its possible outcomes

Exclusion Criteria:

* - Treatment with a laryngeal mask
* If a traumatic extraction is needed, this patient is excluded from the study
* Children who do not meet the inclusion criteria
* Deviation in the pain relief protocol
* Parents/child don't speak Dutch
* Patients with missing data during the procedure/follow-up

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium in the child (flowchart) | 5 minutes after spontaneous eye opening
  to investigate whether the administration of intra-osseous local anaesthesia (Quicksleeper 5, an electronically controlled intra-osseous anaesthesia injection system) to children during general anaesthesia prior to the extraction of a first permanent molar (FPM) has an effect on immediate and later postoperative delirium in the child. Postoperative delirium will be assessed 5 min after spontaneous eye opening using a validated flowchart
Pre- and postoperative pain in the child (Visual Analogue Scale - VAS) | Preoperative: upon arrival at the hospital Postoperative: after 120 minutes
  to investigate whether the administration of intra-osseous local anaesthesia (Quicksleeper 5, an electronically controlled intra-osseous anaesthesia injection system) to children during general anaesthesia prior to the extraction of a first permanent molar (FPM) has an effect on immediate and later postoperative pain in the child. Pre-and postoperative pain will be assessed at a fixed time after the procedure (after 120 minutes) using the validated VAS (Visual Analogue Scale) scale. Upon arrival at the hospital, the preoperative VAS will be taken.
  The scale consists of a line of numbers from 0 (left side of the line) to 10 (right side of the line). The higher the number, the more pain, so a worse outcome.
Pre- and postoperative pain in the child (Face-Legs-Activity-Cry-Consolability Scale) | Preoperative: arrival at the hospital, postoperative: after 10,30,60,120 minutes
  to investigate whether the administration of intra-osseous local anaesthesia (Quicksleeper 5, an electronically controlled intra-osseous anaesthesia injection system) to children during general anaesthesia prior to the extraction of a first permanent molar (FPM) has an effect on immediate and later postoperative pain in the child. Pre-and postoperative pain will be assessed at fixed times after the procedure (after 10/30/60/120 minutes) using the validated FLACC (Face-Legs-Activity-Cry-Consolability Scale) scales. Upon arrival at the hospital, the preoperative FLACC will be taken.
  The scale consists of 5 scores assigned by an observer based on child's behavior/attitude. The sum of these determines the pain. 0 is no pain, 10 is intense pain. The higher the score, the outcome is worse.
Pre- and postoperative anxiety in the child (CFSS-DS - Children's Fear Survey Schedule - Dental Subscale) | Preoperative: upon arrival at the hospital Postoperative: after 120 minutes
  to investigate whether the administration of intra-osseous local anaesthesia (Quicksleeper 5, an electronically controlled intra-osseous anaesthesia injection system) to children during general anaesthesia prior to the extraction of a first permanent molar (FPM) has an effect on immediate and later postoperative anxiety in the child. Postoperative anxiety will be assessed at a fixed time after the procedure (after 120 minutes) using a validated scale (CFSS-DS - Children's Fear Survey Schedule - Dental Subscale). The scale consists of 15 questions with a score from 1 till 5. A score of 15 in total means no anxiety, a higher score means more dental anxiety/fear, so a worse outcome.

SECONDARY OUTCOMES:
presence of postoperative side effects related to local anesthesia | 10 minutes up to 24 hours 10, 30, 60, 120 minutes after waking up (VAS - Visual Analogue Scale, FLACC - Face, Legs, Activity, Cry and Consolability, CFSS-DS- Children's Fear Survey Schedule - Dental Subscale questionnaire). After 24 hours: QoR-15
  the presence of postoperative side effects related to local anesthesia (bite wounds, numbness, postoperative bleeding, vomiting, nausea, etc.) will be evaluated.
  After 24 hours, parents will be asked to complete the Quality of Recovery15 (QoR-15) digitally (qr-code). This is a validated scale.

OTHER OUTCOMES:
Possible influence of the child's gender, site of extraction (maxilla or mandible/left or right) | up to 24 hours
  The investigators will examine whether there is a possible influence of the child's sex and the site of extraction (maxilla or mandible/left or right) on pain and anxiety perception of the child. The Quality of Recovery -15 will be used for this purpose as well as geographical data from the surgical report (was the extracted tooth in the maxilla or mandible, left or right). This questionnaire consists of 15 questions, which are scored from 0 till 10. The higher the score, the better the quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Chloë Sterkens, Principal Investigator — Equal Lifelong Oral Health for All Research Group, Paediatric Dentistry
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The IPD must be shared as anonymized or pseudonymized information. Data transfer must be conducted under Ghent University Hospital conditions, with legal experts drafting and reviewing the agreement (https://hiruz.be/cu/). Additionally, any data containing personal information requires approval from the Ethics Committee before transfer.